CLINICAL TRIAL: NCT06402513
Title: A Phase 1 Study in Healthy Adult Subjects to Evaluate the Pharmacokinetics, Immunogenicity, Safety, and Tolerability of a Ravagalimab Subcutaneous Formulation in a Pre-Filled Syringe
Brief Title: A Study in Healthy Adult Participants to Assess the Pharmacokinetics, Immunogenicity, Safety, and Tolerability of a Ravagalimab Subcutaneous Formulation in a Pre-Filled Syringe
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M24-518
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; Ravagalimab; ABBV-323

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ravagalimab (Experimental): Participants will receive 2 (SC) subcutaneous injections of Ravagalimab via Pre-Filled Syringe at Day 1 and followed for 85 days
  Interventions: Drug: Ravagalimab

INTERVENTIONS:
Drug: Ravagalimab — Subcutaneous Injection
  Other Names: ABBV-323

SUMMARY:
The objective of this study is to assess the pharmacokinetics, immunogenicity, safety, and tolerability, of subcutaneous formulation of ravagalimab in a pre-filled syringe in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) is ≥ 18.0 to ≤ 29.9 kg/m^2 after rounding to the tenth decimal at screening.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead ECG.

Exclusion Criteria:

* History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.
* Participant using any over the counter and/or prescription medication, vitamins and/or herbal supplements, with the exception contraceptives or hormonal replacement therapies for females, on a regular basis.
* History of any clinically significant sensitivity or allergy to any medication or food.
* No prior exposure to ravagalimab
* Participant using any medications, vitamins, and/or herbal supplements within the 2-week period or 5 half-lives (whichever is longer) prior to study drug administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Approximately up to 71 days
  Maximum Observed Plasma Concentration (Cmax)
Time to Maximum Observed Plasma Concentration (Tmax) | Approximately up to 71 days
  Time to Maximum Observed Plasma Concentration (Tmax)
Apparent Terminal Phase Elimination Rate Constant (β) | Approximately up to 71 days
  Apparent Terminal Phase Elimination Rate Constant (β)
The Terminal Phase Elimination Half-Life (t1/2) | Approximately up to 71 days
  The Terminal Phase Elimination Half-Life (t1/2)
The Area Under the Plasma Concentration-Time Curve (AUC) from Time 0 to Time of the Last Measurable Concentration (AUCt) | Approximately up to 71 days
  The Area Under the Plasma Concentration-Time Curve (AUC) from Time 0 to Time of the Last Measurable Concentration (AUCt)
The Area Under the Plasma Concentration-Time Curve (AUC) from Time 0 to Infinity (AUC∞) | Approximately up to 71 days
  The Area Under the Plasma Concentration-Time Curve (AUC) from Time 0 to Infinity (AUC∞)
Number of Anti-drug antibody (ADA) Titers | Approximately up to 71 days
  Incidence of anti-drug antibodies
Number of Participants with Adverse Events | Approximately up to 85 days
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 265325, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-518